CLINICAL TRIAL: NCT04559438
Title: Post-operative Pain Following Glide Path Preparation Using Rotary Neoniti GPS File and Manual K-files in Non-vital Lower Molars: A Randomized Controlled Trial
Brief Title: Post-operative Pain Following Glide Path Preparation Using Rotary Neoniti GPS File and Manual K-files
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Abdel Nour Atallah, Principal investigator, Resident at faculty of dentistry, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENDO 3-3-5
Record Dates: First submitted 2020-09-10; First posted 2020-09-22 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotary Neoniti GPS (Experimental): Glide path preparation using Rotary Neoniti GPS file (Neolix, châtres-la-Forêt, France).
  Interventions: Other: Rotary Neoniti GPS file
- Stainless steel K-files (Active Comparator): Glide path preparation using manual stainless steel K-files #10, #15 (Dentsply Maillefer, Ballaigues, Switzerland).
  Interventions: Other: Manual stainless steel K-files

INTERVENTIONS:
Other: Rotary Neoniti GPS file — Glide path creation will be achieved using Neoniti GPS file (15/.03). The file will be introduced passively inside the canal, in continuous rotation at a constant speed between 300 and 500 rpm and torque of 1.5 N.
  Arms: Rotary Neoniti GPS
Other: Manual stainless steel K-files — Glide path preparation will be done by hand instrumentation using K-files #10 and 15.
  Arms: Stainless steel K-files

SUMMARY:
The aim of this study is to clinically compare the incidence of post-operative pain after using rotary glide path file (Neoniti GPS), on post-operative pain when compared to manual glide path preparation in lower molars with asymptomatic non-vital pulp.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy patients (ASA I or II)
2. Lower permanent molar teeth with:

Asymptomatic non-vital pulps, No response of pulp tissue to cold pulp tester (ethyl chloride spray), with or without periapical lesions.

Exclusion Criteria:

1. Medically compromised patients having significant systemic disorders. (ASA III or IV).
2. History of intolerance to NSAIDS.
3. Patients with two or more adjacent teeth requiring endodontic treatment.
4. TMJ problems, bruxism, clenching or traumatic occlusion.
5. Inability to perceive the given instructions.
6. Teeth with:

Vital pulp tissues. Association with swelling. Acute periapical abscess. Mobility Grade II or III. Pocket depth more than 5mm. Previous root canal therapy. Non-restorability.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain assessed using the Visual Analogue Scale | 6 hours post treatment.
  Intensity of pain after root canal treatment will be recorded by the patient where; "0" = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain.
Postoperative pain assessed using the Visual Analogue Scale | 12 hours post-treatment.
  Intensity of pain after root canal treatment will be recorded by the patient where; "0" = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain.
Postoperative pain assessed using the Visual Analogue Scale | 24 hours post-treatment.
  Intensity of pain after root canal treatment will be recorded by the patient where; "0" = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain.
Postoperative pain assessed using the Visual Analogue Scale | 48 hours post-treatment.
  Intensity of pain after root canal treatment will be recorded by the patient where; "0" = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain.
Postoperative pain assessed using the Visual Analogue Scale | 72 hours post treatment.
  Intensity of pain after root canal treatment will be recorded by the patient where; "0" = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain.

SECONDARY OUTCOMES:
Number of analgesic tablets taken by the patient | Up to 72 hours post treatment.
  Number of analgesic tablets taken by the patient after root canal treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Heba ElFar, Professor, Study Chair — Cairo University (Endodontics Department); Dina Morsy, Lecturer, Study Director — Cairo University (Endodontics Department)
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pasqualini D, Mollo L, Scotti N, Cantatore G, Castellucci A, Migliaretti G, Berutti E. Postoperative pain after manual and mechanical glide path: a randomized clinical trial. J Endod. 2012 Jan;38(1):32-6. doi: 10.1016/j.joen.2011.09.017. Epub 2011 Oct 27. PMID 22152616
- [Background] Keskin C, Sivas Yilmaz O, Inan U, Ozdemir O. Postoperative pain after glide path preparation using manual, reciprocating and continuous rotary instruments: a randomized clinical trial. Int Endod J. 2019 May;52(5):579-587. doi: 10.1111/iej.13053. Epub 2018 Dec 31. PMID 30536837
- [Background] West JD. The endodontic Glidepath: "Secret to rotary safety". Dent Today. 2010 Sep;29(9):86, 88, 90-3. PMID 20973422